CLINICAL TRIAL: NCT00319423
Title: Evaluation of Function and Effect of Exercise Therapy in Patients With Osteoarthritis of the Hip. A Randomized Controlled Trial.
Brief Title: Exercise Therapy and Patient Education for Individuals With Hip Osteoarthritis. a RCT.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03a-2005-NAR
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2006-04

CONDITIONS: Hip Osteoarthritis
Keywords: Hip Osteoarthritis, Exercise therapy, Patient Education
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Patient education (Active Comparator): Patient education according to Klassbo et al 2003
  Interventions: Procedure: Patient education and supervised exercise
- Patient education and supervised exercise (Experimental): Patient education according to Klassbo et al 2003. Supervised exercise containing strengthening, functional and flexibility exercises.
  Interventions: Procedure: Patient education and supervised exercise

INTERVENTIONS:
Procedure: Patient education and supervised exercise — Patient education: 3 sessions Supervised exercise: 2-3 times/week for 12 weeks

SUMMARY:
Aims:

1. Evaluate the effect of an exercise therapy program and patient education, versus patient education only, on hip function among patients with radiologically verified hip OA
2. To identify biomechanical differences during gait, one-leg standing , and two-legged-raise analysis in patients with hip OA following either exercise therapy and patient education program, or a patient education program only.

Main Hypothesis:

Significant improved hip function (WOMAC) will be demonstrated in patients with hip osteoarthritis (OA) (radiographically verified hip OA) following a patient education program and a 12 week exercise therapy program, compared to those only going through a patient education program.

Material and Methods:

110 patients with radiographically verified hip OA will be included in the randomized controlled trial; they will be randomized into:

1. Patient Education, or
2. Patient Education in addition to a supervised exercise program.

The main outcome is:

The Disease Specific WOMAC-Index.

Secondary outcome measures are:

SF-36v2 (quality of life),PASE (activity score), Self-efficacy for pain, muscle strength tests, gait analysis (biomechanical analysis),6 minutes walking test, Åstrand's bike test, range of motion.

Status:

The PhD student is accepted at the University of Oslo,and the study has so far included 17 subjects.

The study will be carried out:

NAR-Orthopedic Centre, Ullevaal University Hospital in collaboration with Diakonhjemmet Hospital and University of Delaware.

The study is included in our research program for active rehabilitation.

DETAILED DESCRIPTION:
Aim 1:

To evaluate the effect of an exercise therapy program for 12 weeks and a patient education program compared to a patient education program only on hip function (WOMAC) in patients with hip osteoarthritis (OA) (radiographically verified hip OA, Harris Hip Score 60-95p, and >3 months of hip pain).

Aim 2:

To identify biomechanical differences during gait analysis in patients with hip OA following either exercise therapy and patient education program, or a patient education program only.

Main hypothesis:

Significant improved hip function (WOMAC) will be demonstrated in patients with hip osteoarthritis following a patients education program with an additionally 12 week exercise therapy program, compared to those only going through a patient education program.

MATERIAL AND METHODS

Design:

A randomized controlled trial.

Inclusion Criteria:

Patients between 40 and 80 years old with uni- or bilateral hip disability not eligible for hip surgery will be recruited from Orthopaedic Centre, Ullevål University Hospital, NIMI, and Diakonhjemmets Sykehus (Hospital), Oslo. Inclusion criteria for all subjects are:

* Harris Hip Score (35) between 60 and 95, and hip pain of more than 3 months. Harris Hip Score (35) of 60 or below are used regularly at our institution as one of the criteria for hip surgery (arthroplasty), therefore Harris Hip Score between 60 and 95 is used as inclusion criteria for the present study population.
* All subjects will have x-ray taken. Those with radiographic verified hip OA will be classifies by an orthopaedic surgeon (LN) according to Danielsson's criteria for radiographic hip OA (34).

One hundred and ten patients with radiographic verified hip OA will be included in the randomized controlled trial

Exclusion Criteria

* Patients will be excluded if they have a history of resent trauma or functional impairment to the lower limbs or diseases which might interfere with participation (rheumatoid arthritis, cancer, osteoporosis, severe back pain, knee OA).
* Patients with co-morbidities not tolerating physical activities will be excluded.

Interventions It is not considered ethically or practically feasible to use a control group receiving no treatment in this study. Hence, both randomized groups will be offered the patient education intervention, and one of the groups will receive exercise therapy in addition.

Patient Education (KLASSBO M, 2003):

All patients with hip disability with or without verified radiographic OA included in the study will receive two individual and three small-group (6-7 patients) sessions lasting one hour each time.

Exercise Protocol:

The exercise protocol includes exercises from former studies on comparable patient populations. The intensity of the strength- and flexibility exercises meets the American College of Sports Medicine's (ACSM) recommendations for developing and maintaining muscular fitness in adults.Patients will be required to exercise for 60 minutes, three days a week for 12 weeks. Patient's attendance to the exercise program (compliance) will be registered by the physical therapists.

Outcome Measurements

Pain and Functional Activity:

The primary (main) outcome measurement will be the self-reported functional outcome measure, the disease-specific questionnaire Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). WOMAC is found to be a valid, reliable and responsive outcome measure in patients with hip OA.

The self-reported Physical Activity Score for the Elderly (PASE) will be used to record the individuals activity level prior to inclusion and at follow-up intervals. Hip pain will be recorded on a visual analogue scale (VAS) rating from 0 to 100 mm; 0 represents "no pain" and 100 represents "as much pain he/she can possibly imagine". The pain will be recorded after the 6 minutes walking test (se below).

Six minutes walking tests (Enright, 2003): Observed functional capacity and cardiovascular fitness will be assessed by a six minute walk test. This test has been reliability estimated for older adults and validated for older adults and individuals with total hip arthroplasty.

Health related quality of life and pain management: Quality of life will be assessed by using the self-administered generic questionnaire 36-item short-form health survey (SF-36) version 2.

Hip Biomechanics:

Gait analysis:

Kinematic data will be collected using Qualisys pro-reflex motion analysis system with eight cameras at a sampling frequency of 240 Hz and synchronized with two force platforms sampling at a rate of 960 Hz (AMTI Model LG6).

Subjects will be instructed to walk along a 17 m walkway in which two force plates are embedded. Speed will be measured by photoelectric beams located 3.06 m apart, midway along the walkway. Eight to ten walking trials will be averaged for each subject. Kinematic and kinetic variables will include hip, knee, and ankle angles and moments, in the sagittal, frontal and transverse planes. The setup and the analysis software that we used are the same as our collaborative group at the University of Delaware use.

Balance(Suni et al. 1998):

Static balance will be tested by one-leg standing. The subject is advised to stand as still as possible and center of pressure will be registered on a force plate (AMTI Model LG6). The test is developed for adults and has been used in several former studies.

Dynamic balance will be registered by the patient performing a two-legged raise from seated position to standing position on the force plate (Mizner &Snyder-Mackler). Center of pressure, kinematic, and kinetic data will be registered.

Muscle strength: Isokinetic muscle strength will be tested in Technogym REV 9000 (Gambettola, Italia) and measured as peak torque at 60°s-1 for hip flexion/extension, knee flexion/extension and ankle flexion/extension. Muscle strength for hip abduction will be conducted isometrically with a dynamometer.

Cardiovascular Fitness (Åstrand & Rodahl, 1986):

will be tested by a sub-maximal bicycle ergometer test according to the method described by Åstrand & Rodahl. The load will be adjusted to each subject. Results will be corrected for age and gender and expressed in ml O2 / kg / min.

Range of motion:

will be registered with a plastic goniometer. Flexion, abduction, and adduction is registered in supine position, with a fixation of the contralateral leg. Internal and external rotation is registered in prone position with fixation over buttocks. Extension is registered according to Thomas test.

Data Collections and Follow-Up In the randomized controlled trial (Aim 1 and 2), data will be collected at inclusion, after the 15 weeks intervention period, and at follow- ups at 6 months, 1 year, and 2 years. Data from all outcome measurements will be collected from all patients at all follow-ups, except for the gait-analysis data (kinematic and kinetic data) (Aim 2). These data will be collected at inclusion and after the intervention period (15 weeks).

Power Calculations:

The WOMAC Index will be the main outcome measurement in the RCT. Power calculations based on a standard deviation of 23 mm, and a minimum clinically important difference of 15 mm between groups calculated that there is a need for 49 patients in each group. To account for possible drop-outs, 110 patients will be included in the RCT.

Blinding:

Personnel responsible for the intervention will not be involved in data collection. Physical therapists collecting data will be blinded for patients' group allocation. A research coordinate person, not involved in any part of the study intervention or data collections, will be responsible for randomization procedures (give subjects information about group allocation)

Statistical Analysis:

Data in the randomized controlled trial will be analyzed both according to the intention to treat principles and additional analysis for the compliers adhering to the exercise protocol at a cut-off value of 24 or more training sessions.

Registration of Complications, Drop-Outs and Compliance:

Complications and drop-outs will be registered by persons responsible for data collection. There will be used intention to treat analysis. Compliance to the patient education and the exercise protocol will be registered by the physical therapists responsible for the treatment.

Ethics:

All patients and control subjects will receive written and oral information about the study and sign an informed consent before inclusion. The project will be performed according to recommendations of the Helsinki Declaration. Approval is obtained from the Regional Committee of Medical Research Ethics.

ELIGIBILITY:
Inclusion Criteria:

* Between 40 and 80 years old with uni- or bilateral hip disability
* Harris Hip Score (36) between 60 and 95. Harris Hip score (0-100 points) is widely used as an assessment of hip function in patients with hip OA. Harris Hip Score of 60 or below are used regularly at our institution as one of the criteria for hip surgery (arthroplasty).
* Patients will be included if they have more than 3 months of hip pain.
* Patients with radiographic verified hip OA (Danielson's criteria for radiographic OA: Danielsson's criteria for minimal joint space: < 4 mm < 70 years, < 3 mm ≥ 70 years, or 1 mm difference between hips).

Exclusion Criteria:

* Patients have a history of resent trauma or functional impairment to the lower limbs or diseases which might interfere with participation (rheumatoid arthritis, cancer, osteoporosis, severe back pain, knee OA).
* Patients with co-morbidities not tolerating physical activities

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2005-04; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 0, 4, 10, 16 months

SECONDARY OUTCOMES:
SF-36 (quality of life) | 0, 4, 10, 16 months
PASE (activity score) | 0, 4, 10, 16 months
Self-efficacy for pain | 0, 4, 10, 16 months
Muscle strength tests | 0, 4, 10 months
Gait analysis (biomechanical analysis) | 0, 4 months
6 minute walk test | 0, 4, 10 months
Åstrand's bike test | 0, 4, 10 months
Range of motion | 0, 4, 10 months

CONTACTS AND LOCATIONS:
Overall Officials: May Arna Risberg, PT, PhD, Principal Investigator — NAR- Orthopedic Centre, Ullevål University Hospital
Locations (1):
- NAR-Orthopedic Centre, Ullevål University Hospital & NIMI, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Eitzen I, Fernandes L, Kallerud H, Nordsletten L, Knarr B, Risberg MA. Gait Characteristics, Symptoms, and Function in Persons With Hip Osteoarthritis: A Longitudinal Study With 6 to 7 Years of Follow-up. J Orthop Sports Phys Ther. 2015 Jul;45(7):539-49. doi: 10.2519/jospt.2015.5441. Epub 2015 May 21. PMID 25996360
- [Derived] Eitzen I, Fernandes L, Nordsletten L, Risberg MA. No effects of a 12-week supervised exercise therapy program on gait in patients with mild to moderate osteoarthritis: a secondary analysis of a randomized trial. J Negat Results Biomed. 2015 Mar 5;14:5. doi: 10.1186/s12952-015-0023-y. PMID 25886499
- [Derived] Svege I, Nordsletten L, Fernandes L, Risberg MA. Exercise therapy may postpone total hip replacement surgery in patients with hip osteoarthritis: a long-term follow-up of a randomised trial. Ann Rheum Dis. 2015 Jan;74(1):164-9. doi: 10.1136/annrheumdis-2013-203628. Epub 2013 Nov 19. PMID 24255546
- [Derived] Eitzen I, Fernandes L, Nordsletten L, Risberg MA. Sagittal plane gait characteristics in hip osteoarthritis patients with mild to moderate symptoms compared to healthy controls: a cross-sectional study. BMC Musculoskelet Disord. 2012 Dec 20;13:258. doi: 10.1186/1471-2474-13-258. PMID 23256709
- [Derived] Fernandes L, Storheim K, Sandvik L, Nordsletten L, Risberg MA. Efficacy of patient education and supervised exercise vs patient education alone in patients with hip osteoarthritis: a single blind randomized clinical trial. Osteoarthritis Cartilage. 2010 Oct;18(10):1237-43. doi: 10.1016/j.joca.2010.05.015. Epub 2010 Jul 13. PMID 20633669